CLINICAL TRIAL: NCT05207189
Title: Phase II Study Evaluating the Treatment of Women Urinary Incontinence by Suburethral Slings; UVT Allograft; in Patients Presenting With Complication of the Synthetic Sling Treatment
Brief Title: Biological Sling Allograft (UVT) for the Treatment of Urinary Incontinence in Women Presenting With Synthetic Sling Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVT-TBF1; 2020-A02983-36 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-12-28; First posted 2022-01-26 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Female Stress Incontinence; Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UVT (Experimental): Biological sling used as a replacement of the synthetic sling.
  Interventions: Biological: UVT

INTERVENTIONS:
Biological: UVT — Chemically-treated, viro-inactivated, freeze-dried and irradiated umbilical vein allograft placed in replacement of a failed synthetic sling during a surgical act performed by the investigator.

SUMMARY:
The purpose of this open, multi center trial is to evaluate a new biological replacement for synthetic slings in the treatment of female stress urinary incontinence.

DETAILED DESCRIPTION:
It was estimated that more than 9 million French people are affected by urinary incontinence, of which 1% are treated surgically. Indeed, if medical treatment or rehabilitation fails, surgical treatment must be considered. Sling implantation is a commonly used surgical technique to treat stress urinary incontinence as it allows for a reduction in surgery time and morbidity and can be placed under local anesthesia. However, the risk of complications associated with the use of synthetic products is high and contributes to the recent decline of popularity of synthetic slings. As the demand for incontinence treatment remains high, fascia autograft surgeries are being proposed, even though they require an additional surgical procedure and expose the patient to complications at the donor site of the graft.

The study product aims to address the growing need for a safer but equally effective implant to avoid autografting while keeping the standard surgical technique.

The aim of this exploratory study is to evaluate a biological sling replacement to failed synthetic slings in the treatment of female stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women over 40 years of age and under 75 years of age.
* Failure of primary surgical technique with synthetic sling requiring its removal due to complications such as vaginal exposure or urinal tract erosion.
* Inclusion more than 3 months after primary surgery.
* Any fistula or abnormality of the urinary tract, any erosion or complication due to the synthetic sling placement must be repaired during surgery. In case of persistence of complication or limited possibility to insert the UVT due to major vesical or urethral lesion, the patient will not be included.
* Patients with controlled urinal tract infections.
* Patients who received the study information and provided consent.
* Patients who are members or the beneficiary of a national health insurance plan.

Exclusion Criteria:

* Breast feeding women or women without effective contraception. In absence of effective contraception, a pregnancy test followed by an effective contraception are mandatories for non-menopausal women.
* Patients with mild cases treated by physiotherapy and pelvic floor exercises for urinary incontinence or without surgical complications.
* Patients with current urinary infection, severe anemia or other pathologies that counter-indicate surgery.
* Cystocele and rectocele not treated during the surgery.
* Persons under guardianship or confined by a judicial or administrative decision.
* Patients unable to have discernment for rehabilitation, unable to perform follow-up or unable to provide their consent.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
No major signs of incontinence | 6 months
  Use of less than 2 pads a day
No complication related to investigational product | 6 months
  Evaluation of urinary retention, dysuria, local inflammation, irritation of suture and suspension areas, and other indirect symptoms

SECONDARY OUTCOMES:
Decrease of the signs of complications of the first surgery | 15 days, 6 weeks, 3 months, 6 months, 12 months
  Monitoring of urinary retention, dysuria, local inflammation, irritation of suture and suspension areas, and other indirect symptoms
Decrease of pain and analgesic consumption | 15 days, 6 weeks, 3 months, 6 months, 12 months
  Pain evaluated from 0: no pain to 10: worst imaginable pain on visual analog scale (VAS)
Progressive recuperation of continence | 15 days, 6 weeks, 3 months, 6 months, 12 months
  Continence evaluated by uroflow test and 3-day voiding diary
Decrease of Urinary Incontinence (UI) severity | 6 weeks, 3 months, 6 months, 12 months
  Decrease in the score of the International Consultation on Incontinence Questionnaire - Urinary Incontinence - Short Form (ICIQ-UI-SF) (0 = no UI, 21 = very severe UI)
Decrease of distress caused by UI symptoms | 6 weeks, 3 months, 6 months, 12 months
  Decrease of the Urogenital Distress Inventory (UDI-6) score (0 = no distress caused by UI symptoms, 100 = highest possible distress cause by UI symptoms)
Improvement of health-related quality of life | 6 weeks, 3 months, 6 months, 12 months
  Decrease of the Incontinence Impact Questionnaire (IIQ-7) score (0 = no impact of UI on health-related quality of life, 100 = highest possible impact of UI on health-related quality of life)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôtel-Dieu, CHU de Nantes, Nantes
  - Hôpital de la Pitié-Salpêtrière, Assistance Publique des Hôpitaux de Paris, Paris
  - Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No